CLINICAL TRIAL: NCT06617013
Title: Characteristics of Gastroesophageal Reflux in Children With Cystic Fibrosis
Brief Title: GERD in Children With Cystic Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00115374
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: GERD in Children; Cystic Fibrosis in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child with cystic fibrosis (CF) on GERD therapy without severe GERD (Experimental): The GSAS will be completed at baseline, GERD therapy will be discontinued, and GSAS will be repeated 12 weeks later.
  Interventions: Other: Discontinuation of GERD therapy
- Child with cystic fibrosis (CF) (No Intervention): The GSAS will be completed at baseline.

INTERVENTIONS:
Other: Discontinuation of GERD therapy — GERD therapy will be discontinued at time of enrollment.
  Arms: Child with cystic fibrosis (CF) on GERD therapy without severe GERD

SUMMARY:
The purpose of this study is to evaluate the prevalence of gastroesophageal reflux disease (GERD) symptoms in pediatric patients with cystic fibrosis using the Gastroesophageal Symptom Assessment Scale (GSAS) and the impact of stopping anti-GERD therapy on the GERD symptoms reported.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-18 years of age with a confirmed CF diagnosis by either a positive sweat test or 2 disease causing CFTR mutations.
* Signed consent

Exclusion Criteria:

* Declining to participate in the study or sign consent
* History of severe GERD per gastroenterology diagnosis and documentation
* GSAS score >80

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean GSAS score (only if GERD medication discontinued) | baseline and 12 weeks
  The Gastroesophageal Reflux Disease Symptom Assessment Scale (GSAS) is a 15-item tool validated in children in assessing gastroesophageal reflux disease-related symptoms. The GSAS ranges from 0 to 490, with a higher score representing worse GERD symptoms, and a score ≥ 15 reflects significant GERD symptoms.
Mean GSAS score in children with CF on GERD therapy | Baseline
  GSAS ranges from 0 to 490, with a higher score representing worse GERD symptoms, and a score ≥ 15 reflects significant GERD symptoms. A value of 80 will be used as a maximum cut-off for mild symptoms as this was 2 SD from the mean GSAS for children without baseline GERD.
Mean GSAS score in children with CF not on GERD therapy | Baseline
  GSAS ranges from 0 to 490, with a higher score representing worse GERD symptoms, and a score ≥ 15 reflects significant GERD symptoms. A value of 80 will be used as a maximum cut-off for mild symptoms as this was 2 SD from the mean GSAS for children without baseline GERD.

CONTACTS AND LOCATIONS:
Overall Officials: Shatha Yousef, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No